CLINICAL TRIAL: NCT07251387
Title: Test-retest Fidelity of a Tool for Calculation of Muscle Synergies
Brief Title: Muscle Synergies in Pain and Pain Anticipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universite de Picardie Jules Verne (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Jennifer Burgos Tirado, Researcher - Ph.D student, Universite de Picardie Jules Verne
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-5551-1H
Record Dates: First submitted 2025-09-22; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pain; Nocebo Effect; Pain Anticipation
Keywords: Nocebo effect; Pain anticipation; Pain; Gait; Motricity; Muscle synergies
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware that a cream applied to them (neutral cream) does not produce any pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prior Experience Group (Experimental): Participants in this arm have experienced capsaicin cream before and will be given a neutral cream. They will be told that the cream contains capsaicin and will cause pain.
  Interventions: Other: Pain expectation conditioning; Other: Gait assesment
- Control Group (Sham Comparator): Pariticpants in this arm have never experienced capsaicin cream before and will be given a neutral cream. They will be told that the cream contains capsaicin and will cause pain.
  Interventions: Other: Pain expectation conditioning; Other: Gait assesment

INTERVENTIONS:
Other: Pain expectation conditioning — Participants receive a neutral cream with no real harmful effects with verbal and behavioral suggestions that it may cause localized pain. Researchers wear gloves during application and emphasize the potential discomfort, stating effects may intensify with movement.
Other: Gait assesment — Gait will be assessed both before and after cream application. Each assessment will consist of walking on a treadmill at varying speeds while physiological data (EMG) is recorded. Identical questionnaires (VAS, TAMPA, and PCS) will be administered immediately following the first gait assessment.

SUMMARY:
This study investigates how the anticipation of pain affects muscle synergies. Two groups will be compared: an experimental group, who first experience actual pain from capsaicin cream and are then presented with a harmless cream deceptively labeled as capsaicin, against a control group, who are presented with a harmless cream labeled as potentially painful, without any prior painful experience. The changes in muscle synergies will be measured during walking tasks.

DETAILED DESCRIPTION:
Participants will be recruited through university announcements. Eligibility will be determined by a screening process that assesses prior experience with capsaicin cream. Healthy adults aged 18-35 who meet the inclusion criteria will be enrolled and assigned to one of two groups based on their screening responses:

1. Experimental Group ("Prior Experience"): Individuals who report a prior painful experience with capsaicin cream.
2. Control Group ("No Prior Experience"): Individuals who report no prior experience with capsaicin cream.

All participants will take part in a single experimental session. Both groups will receive identical negative verbal suggestions indicating that a neutral, harmless cream is a potent capsaicin formulation likely to cause pain.

Participants will complete a walking assessment on a treadmill. The speed will be incrementally increased from 0.8 m/s to 1.1 m/s. Throughout this task, muscle activity will be recorded via electromyography (EMG), and ground reaction forces will be captured by force platforms embedded in the treadmill.

Following the initial walk, participants will complete a set of standardized questionnaires to establish baseline scores for pain perception (Visual Analog Scale, VAS), fear of movement (Tampa Scale of Kinesiophobia, TSK), and pain catastrophizing (Pain Catastrophizing Scale, PCS).

The neutral cream will be applied to the knee, specifically in the area between the lateral epicondyles of the femur, in a 4 cm wide band. Participants will immediately fill out the VAS to report any pain sensations. The walking assessment is repeated, measuring the same physiological signals (EMG and ground reaction forces).

The primary objective is to determine whether a prior painful experience with capsaicin causes individuals to generalize that pain memory to a neutral sensation, leading to different outcomes than in those who only have a negative expectation. We will specifically investigate the magnitude of this effect on muscle synergies and ground reaction forces.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years old
* Healthy participant with no self-reported diagnosed neurological, musculoskeletal, or cardiovascular disorders
* Body Mass Index (BMI) < 30
* Ability to walk unaided for at least 10 minutes without major physical limitations

Exclusion Criteria:

* Presence of pain at the time of testing
* Self-reported diagnosed condition affecting mobility
* Known allergy to any component of the study cream
* Allergy to EMG electrode adhesives
* Inability to stand unassisted for more than 1 minute
* Inability to walk/run at the required speed and distance
* Weight exceeding 150 kg (due to treadmill limitations)
* Recent intake (prior intervention) of:
* Analgesics (within 6 hours)
* Cigarettes (within 6 hours)
* Caffeine (within 2 hours)
* Skin lesions at the cream application site
* Pregnancy
* Failure to understand instructions
* Daytime pain reported by participant on day of experimentation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of muscle synergies derived by non-negative matrix factorization | Before intervention, after intervention (10 minutes after cream application)
  Changes in the activation of the muscle synergies during the gait cycle.
Changes in Muscle Synergy Composition derived by non-negative matrix factorization. | Before intervention, after intervention (10 minutes after cream application)
  Changes in the composition of muscle synergies (i.e., the individuals muscles that comform one muscle synergy)

SECONDARY OUTCOMES:
Pain Catastrophizing (PCS) | Before intervention.
  Pain Catastrophizing Scale total score (0-52). Users rate 13 statements on a scale from 0 (not at all) to 4 (all the time).
Tampa Scale for Kinesiophobia (TSK) | Before intervention.
  Tampa Scale of Kinesiophobia total score (17-68). Users rate 17 statements in a scale from 1 (Strongly disagree) to 4 (Strongly agree).
Self-Reported Pain (VAS) | Before cream application of the cream (pre-intervention) and 10 minutes after cream application (post-intervention).
  Visual Analog Scale (0-100 mm) for immediate pain intensity, where 0 = "No pain" and 100 = "Worst pain imaginable."
Force reactions | Before intervention, after intervention (10 minutes after cream application)
  Ground reaction forces obtained by the instrumented treadmill.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lelard, PhD, HDR, Study Director — Lecturer; Maryne Cozette, PhD, Lecturer, Study Director — Lecturer; Guillaume Léonard, PhD, Lecturer, Study Director — Lecturer
Locations (2):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Canada
- Université de Picardie Jules Verne, Amiens, France

IPD SHARING:
Plan to Share IPD: No
Participants consented to data use only for this specific study under approved protocols.
  Regulations prohibit broad sharing of pseudonymized sensor/video data that could potentially be re-identified (e.g., physical features in GoPro videos, unique gait patterns).

REFERENCES:
- [Background] Nishi Y, Osumi M, Sumitani M, Yozu A, Morioka S. Kinematic changes in goal-directed movements in a fear-conditioning paradigm. Sci Rep. 2021 May 27;11(1):11162. doi: 10.1038/s41598-021-90518-7. PMID 34045515
- [Background] Horvath A, Koteles F, Szabo A. Nocebo effects on motor performance: A systematic literature review. Scand J Psychol. 2021 Oct;62(5):665-674. doi: 10.1111/sjop.12753. Epub 2021 Jun 18. PMID 34145580
- [Background] Escalona MJ, Bourbonnais D, Goyette M, Le Flem D, Duclos C, Gagnon DH. Effects of Varying Overground Walking Speeds on Lower-Extremity Muscle Synergies in Healthy Individuals. Motor Control. 2021 Jan 27;25(2):234-251. doi: 10.1123/mc.2020-0008. PMID 33503586